CLINICAL TRIAL: NCT01204645
Title: Stockholmheartbank and Karolinska Cardiorenal Theme-centre, From Genome to Clinical Practice in Patients With Acute Coronary Syndrome and Impaired Kidney Function
Brief Title: Karolinska Cardiorenal Theme-centre and StockholmHeartbank
Acronym: KKT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Danderyd Hospital (Other)
Collaborators: Region Stockholm (Other Government); Karolinska Institutet (Other); Uppsala University (Other); Lund University (Other); Stockholm South General Hospital (Other); Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Jonas Spaak, MD PhD, Danderyd Hospital
Other Study IDs: KKT
Record Dates: First submitted 2010-09-16; First posted 2010-09-17 (Estimated); Last update posted 2017-06-15 (Actual); Status verified 2017-06

CONDITIONS: Chronic Kidney Disease; Chronic Renal Failure; Acute Coronary Syndrome; Ischemic Heart Disease; Myocardial Infarction
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic; Acute Coronary Syndrome; Myocardial Ischemia; Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and plasma.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Acute Coronary Syndrome (ACS): Continuous inclusion at emergency hospitals of patients with acute coronary syndrome (according to ESC/AHA definitions)
- Follow up: Patients included at 6 or 12 months follow-up visit after an acute coronary event.
- Coronary: Patients included when undergoing an coronary angiography for suspected or confirmed coronary heart disease

SUMMARY:
Chronic kidney disease (CKD) affects 10-18% of the adult population and is becoming recognized as one of the most serious disorders causing increased risk for cardiovascular disease and death. In patients with ischemic heart disease 26% have increased creatinine, which rises to 40% if patients also have diabetes mellitus. Risk increases as renal function diminishes, and just slowing the rate of decline in renal function would have a tremendous impact on health and morbidity. This association is commonly termed the Cardiorenal Syndrome, though it is caused by a much more complex interplay between major pathogenetic pathways such as glucose metabolism and diabetes, systemic and tissue inflammation, tissue metabolism, coagulation, mineral metabolism, sympathetic activation, renin-angiotensin-aldosterone system activation, endothelial dysfunction, lipid metabolism, fetal programming etc.

Karolinska Institutet recently merged basic and clinical researchers in all these fields, creating a Karolinska Kardiorenal Theme Centre; ultimately aiming to explore the syndrome and provide improved care for the individual patient.

The investigators road to success:

* Creating a Biobank (blood, DNA, plasma) from the majority of all hosptalized patients with ACS in Stockholm county - Stockholmheartbank.
* This Theme Center include all teaching hospitals associated with Karolinska Institutet; Danderyd University Hospital, Karolinska University Hospital and Södersjukhuset University Hospital. Together theses hospitals serve as emergency hospitals for 1.9 million people. The investigators are aiming at creating a biobank from all patients admitted for an acute coronary event (about 2.300/yr), which is a unique asset for molecular and genetic research as well as observational and intervention studies.
* The investigators have access to the National registry with 100% coverage, that contains data on all patients admitted to Stockholms coronary care units since 1995.
* To ensure translation in to clinical practice, most of the researchers are also MD:s, and several are clinically active.
* The clinical network facilitates the development of novel therapies and translational research.
* Steering groups for Education and a Clinical Practice implementation program.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to one of the four major emergency hospitals in Stockholm, for an acute coronary event.
* All patients admitted to one of the four major emergency hospitals in Stockholm, for an elective coronary angiography

Exclusion Criteria:

* Severe hemodynamic instability with the need of inotropic therapy and at the same time anemia with haemoglobin <1.1 g/dL

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 1. All patients admitted to one of the four major emergency hospitals in Stockholm, for an acute coronary event.
  2. All patients admitted to one of the four major emergency hospitals in Stockholm, for an elective coronary angiography
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2010-05; Primary Completion 2022-05 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Composite | 1 year
  Combined endpoint of death, new cardiovascular event or dialysis.

SECONDARY OUTCOMES:
Renal function decline | 5 year
Vascular function | 1 year
  Vascular function assessed by arterial stiffness, microcirculation by Laser-Doppler

CONTACTS AND LOCATIONS:
Overall Officials: Jonas Spaak, MD PhD, Study Director — Karolinska Institutet and Danderyd University Hospital
Locations (1):
- Danderyd University Hospital, Stockholm, Sweden